CLINICAL TRIAL: NCT03840408
Title: Prospective Clinical Study of Mitochondria-targeted System Therapy Combined With Radiofrequency Ablation for Early-stage Non-small Cell Lung Cancer
Brief Title: Mitochondria-targeted System Therapy Combined With Radiofrequency Ablation for Early-stage Non-small Cell Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ming Li, Associate senior doctor, Shanghai 10th People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Shanghai
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiofrequency Ablation; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mitochondrial therapy with radiofrequency ablation (Experimental)
  Interventions: Other: Mitochondria-targeted System Therapy Combined With Radiofrequency Ablation
- Surgery (Active Comparator)
  Interventions: Procedure: Surgery

INTERVENTIONS:
Other: Mitochondria-targeted System Therapy Combined With Radiofrequency Ablation — Patients will be treated with mitochondria-targeted system therapy and radiofrequency ablation in the primary tumor sites
  Arms: Mitochondrial therapy with radiofrequency ablation
Procedure: Surgery — Patients will be treated with surgery
  Arms: Surgery

SUMMARY:
Lung cancer is the leading cause of cancer related mortality. Among them, non small cell lung cancer accounts for 85%. Only part of patients could be treated with radical surgery. Mitochondria-targeted system therapy combined with radiofrequency ablation could be an alternative treatment. Small sample clinical cases verified that this therapy could be an efficacy and safe treatment in a short period. The primary aim of this trial is to determine if the efficacy of mitochondria-targeted system therapy combined with radiofrequency ablation is comparable to that of standard surgical interventions for patients with non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* The patient can understand and voluntarily join the study, sign the informed consent form, and the compliance is good.
* Patients with single nodule.
* Before IIB period according to the eighth edition of the TNM staging period.
* No mediastinal lymph node metastasis.
* No prior anticancer treatments including surgery, radiation,chemotherapy or local treatments.
* Eastern Cooperative Oncology Group performance status of 0 to 1
* Sufficient organ functions

Exclusion Criteria:

* Active bacterial or fungous infection.
* Simultaneous or metachronous (within the past 5 years) double cancers.
* Patients with contraindications to radiofrequency ablation and inability to complete treatment;
* Women during pregnancy or breast-feeding.
* Uncontrollable diabetes mellitus.
* Patients with severe heart, lung, kidney disease or other systemic diseases who have been judged to have a severe impact on survival or who are pre-assessed to be unable to tolerate thoracoscopic surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1753 (Estimated)
Dates: Start 2019-01-31 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | From the date of randomization until the date of first documented progression，assessed up to 60 months

SECONDARY OUTCOMES:
Overall survival | From the date of randomization until the date of death from any cause，assessed up to 60 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai 10th People's Hospital, Shanghai, Shanghai Municipality, China